CLINICAL TRIAL: NCT01512745
Title: A Randomized, Double Blinded, Placebo Controlled Multicenter Phase III Study of Apatinib Mesylate Tablets in the Treatment of Advanced or Metastatic Gastric Cancer
Brief Title: Phase III Study of Apatinib Tablets in the Treatment of Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Fudan University (Other); The 81 Hospital of PLA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HENGRUI 20101208
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2015-04

CONDITIONS: Advanced or Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- apatinib (Experimental)
  Interventions: Drug: apatinib
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: apatinib — apatinib 850 mg qd p.o. until disease progression or intolerable toxicity or patients withdrawal of consent
  Arms: apatinib
Drug: placebo — placebo qd p.o. until disease progression or intolerable toxicity or patients withdrawal of consent
  Arms: placebo

SUMMARY:
Apatinib is a tyrosin-inhibitor agent targeting at vascular endothelial growth factor receptor (VEGFR), and it's anti-angiogenesis effect has been viewed in preclinical tests. The investigators' phase I study has shown that the drug's toxicity is manageable and the maximum tolerable daily dose is 850 mg. The purpose of this study is to determine whether apatinib can improve progression free survival or overall survival compared with placebo in patients with metastatic gastric carcinoma who failed two lines of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age
* Histological confirmed advanced or metastatic adenocarcinoma of the stomach
* Have failed for at least 2 lines of chemotherapy
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1 within 1 week before randomization.
* At least one measurable lesion beyond stomach (larger than 10 mm in diameter by spiral CT scan)
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin
* More than 4 weeks for operation or radiotherapy
* More than 4 weeks for cytotoxic agents or growth inhibitors
* Adequate hepatic, renal, heart, and hematologic functions (HB ≥ 90g/L,platelets > 80 ×10 E+9/L, neutrophil > 1.5 × 10 E+9/L, serum creatinine ≤ 1× upper limit of normal(ULN), bilirubin < 1.25× ULN, and serum transaminase ≤ 2.5× ULN).

Exclusion Criteria:

* Pregnant or lactating women
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg).
* Any factors that influence the usage of oral administration; Evidence of Central Nerves System(CNS) metastasis
* Intercurrence with one of the following: coronary artery disease, arrhythmia ,heart failure and proteinuria ≥ (+)
* International Normalize Ratio (INR) > 1.5 and activated partial thromboplastin time（APPT） > 1.5 × ULN
* Abuse of alcohol or drugs
* Certain possibility of gastric or intestine hemorrhage
* Less than 4 weeks from the last clinical trial
* Prior VEGFR inhibitor treatment
* Disability of serious uncontrolled intercurrence infection Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, Pneumoconiosis, radiation pneumonitis, drug-related pneumonia, Pulmonary function damaged seriously etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, PHD, Principal Investigator — Fudan University; Shukui Qin, MD, Principal Investigator — The 81 Hospital of PLA
Locations (2):
- China (2):
  - The 81 Hosiptal of PLA, Nanjing, Jiangsu
  - Fudan University cancer hospital, Shanghai, Shanghai Municipality

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apatinib | Placebo
Started | 176 | 91
Completed | 136 | 71
Not Completed | 40 | 20
Not completed — Adverse Event | 22 | 3
Not completed — Death | 9 | 13
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 4 | 0
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: 5 participants in the apatinib group and 1 in the placebo group withdrew from the study before receiving the assigned treatments.As a result,267 randomly assigned participants were included in Full Analysis Set （FAS），with 176 assigned to the apatinib group and 91 assigned to the placeo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apatinib | Placebo | Total
Number analyzed (Participants) | 176 | 91 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.01 (9.92) | 56.08 (9.74) | 55.37 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 22 | 66
  Male | 132 | 69 | 201

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival(PFS)
Description: Progression free survival of All the Evaluable Participants.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of diameters of target lesions, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 176 | 91
month | 2.6 [2.0 to 2.9] | 1.8 [1.4 to 1.9]

2. Primary Outcome: Overall Survival(OS)
Description: Overall Survival of the Participants
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 176 | 91
month | 6.5 [4.8 to 7.6] | 4.7 [3.6 to 5.4]

3. Secondary Outcome: Disease Control Rate(DCR)
Description: Disease control is defined as the proportion of patients who had a best response rating of complete response, partial response, or stable disease, and lasted at least 4 weeks.
Time Frame: 30 months
Measure: Number; unit: percentage of participants
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 176 | 91
percentage of participants | 42.05 | 8.79

4. Secondary Outcome: Objective Response Rate(ORR)
Description: Objective Response Rate is defined as the proportion of patients with complete response(CR) or partial response(PR)
Time Frame: 30 months
Measure: Number; unit: percentage of participants
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 176 | 91
percentage of participants | 2.84 | 0.00

5. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: 30 months
Measure: Number; unit: percentage of participants
Arm/Group | Apatinib | Placebo
Number analyzed (Participants) | 176 | 91
percentage of participants | 98.30 | 90.11

ADVERSE EVENTS:
Arm/Group | Apatinib | Placebo
Serious Adverse Events (participants affected / at risk) | 6/176 | 6/91
Other Adverse Events (participants affected / at risk) | 173/176 | 82/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apatinib (N=176) | Placebo (N=91)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 5 (5) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apatinib (N=176) | Placebo (N=91)
proteinuria (Renal and urinary disorders) | 84 (84) | 15 (15)
hypertension (Vascular disorders) | 62 (62) | 5 (5)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 49 (49) | 2 (2)
elevated transaminase (Hepatobiliary disorders) | 49 (49) | 20 (20)
hyperbilirubinemia (Hepatobiliary disorders) | 43 (43) | 13 (13)
bleeding (Blood and lymphatic system disorders) | 35 (35) | 22 (22)
fatigue (General disorders) | 36 (36) | 13 (13)
ALP increased (Hepatobiliary disorders) | 35 (35) | 14 (14)
elevated GGT (Hepatobiliary disorders) | 29 (29) | 15 (15)
abdominal pain (Gastrointestinal disorders) | 28 (28) | 16 (16)
decreased appetite (Metabolism and nutrition disorders) | 26 (26) | 8 (8)
hypoproteinemia (Metabolism and nutrition disorders) | 23 (23) | 8 (8)
diarrhea (Gastrointestinal disorders) | 20 (20) | 3 (3)
elevated LDH (Investigations) | 18 (18) | 12 (12)
leukopenia (Blood and lymphatic system disorders) | 71 (71) | 8 (8)
neutropenia (Blood and lymphatic system disorders) | 66 (66) | 9 (9)
anemia (Blood and lymphatic system disorders) | 44 (44) | 22 (22)
thrombocytopenia (Blood and lymphatic system disorders) | 44 (44) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other